CLINICAL TRIAL: NCT02751281
Title: Comparing Pneumatic Versus Ultra-sonic Percutaneous Nephrolithotomy in Large Kidney Stones
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Collaborators: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hamidreza Shemshaki, Dr, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASD-100
Record Dates: First submitted 2016-04-18; First posted 2016-04-26 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Kidney Stone
Keywords: pneumatic; ultra-sonic; percutaneous nephrolithotomy
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pneumatic percutaneous nephrolithotomy (Active Comparator): pneumatic percutaneous nephrolithotomy is type of surgery in treatment of kidney stone
  Interventions: Procedure: Pneumatic percutaneous nephrolithotomy
- Ultra-sonic percutaneous nephrolithotomy (Active Comparator): Ultra-sonic percutaneous nephrolithotomy is type of surgery in treatment of kidney stone
  Interventions: Procedure: Ultra-sonic percutaneous nephrolithotomy

INTERVENTIONS:
Procedure: Pneumatic percutaneous nephrolithotomy — Pneumatic percutaneous nephrolithotomy is type of surgery that we use pneumatic lithotripter to treat kidney stone
  Arms: pneumatic percutaneous nephrolithotomy
Procedure: Ultra-sonic percutaneous nephrolithotomy — Ultra-sonic percutaneous nephrolithotomy is type of surgery that we use ultra-sonic lithotripter to treat kidney stone
  Arms: Ultra-sonic percutaneous nephrolithotomy

SUMMARY:
The purpose of this study is to determine which type of percutaneous nephrolithotomy is better in large kidney stones

DETAILED DESCRIPTION:
While there are several retrospective studies evaluating the efficacy of different lithotripter in percutaneous nephrolithotomy, there are few prospective studies in this regard. This study was designed to compare the efficacy and safety of Ultrasonic versus pneumatic percutaneous nephrolithotomy in treatment of large kidney stones.

ELIGIBILITY:
Inclusion Criteria:

- patients with >2cm kidney stone

Exclusion Criteria:

* Pregnant women
* patients with coagulopathies
* patients with scattered stones who needed several accesses

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2014-12; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
stone free rate | 3 months after surgery

SECONDARY OUTCOMES:
hemoglobin loss | 2 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Nasser Simforoosh, Prof, Study Chair — Shahid Beheshty University of Medical Sciences

IPD SHARING:
Plan to Share IPD: Undecided